CLINICAL TRIAL: NCT01467479
Title: An Open Label,Phase 3 Study of Telaprevir in Combination With Peginterferon Alfa 2a (Pegasys®) and Ribavirin (Copegus®) in Subjects Coinfected With Genotype 1 Hepatitis C Virus and Human Immunodeficiency Virus Type 1(HCV/HIV-1)
Brief Title: A Study to Treat Subjects With Telaprevir, Ribavirin, and Peginterferon Who Are Coinfected With HIV and Hepatitis C Virus (HCV)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: It was decided by Sponsor on 13 January 2014 to terminate study early at primary efficacy endpoint as part of a decision to modify drug development plan.
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX11-950-115
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — telaprevir; Ribavirin; peginterferon alfa-2a; Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- T/PR + HAART Regimen (ATV/r-Based) (Experimental): Participants who were receiving atazanavir/ritonavir (ATV/r) based highly active antiretroviral therapy (HAART) at baseline, received Telaprevir (T)1125 milligram (mg) tablet twice daily for 12 weeks in combination with pegylated interferon alfa 2a (P) (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (R) (RBV) tablet orally twice daily at a dose of 800 milligram per day (mg/day) for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Biological: Pegylated Interferon Alfa-2a; Drug: Highly Active Antiretroviral Therapy (HAART)
- T/PR + HAART Regimen (EFV-Based) (Experimental): Participants who were receiving efavirenz (EFV) based highly active antiretroviral therapy (HAART) at baseline, received Telaprevir (T)1125 milligram (mg) tablet three times a day for 12 weeks in combination with pegylated interferon alfa 2a (P) (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (R) (RBV) tablet orally twice daily at a dose of 800 milligram per day (mg/day) for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Biological: Pegylated Interferon Alfa-2a; Drug: Highly Active Antiretroviral Therapy (HAART)
- T/PR + HAART Regimen (RAL-Based) (Experimental): Participants who were receiving raltegravir (RAL) based highly active antiretroviral therapy (HAART) at baseline, received Telaprevir (T)1125 milligram (mg) tablet twice daily for 12 weeks in combination with pegylated interferon alfa 2a (P) (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (R) (RBV) tablet orally twice daily at a dose of 800 milligram per day (mg/day) for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
  Interventions: Drug: Telaprevir; Drug: Ribavirin; Biological: Pegylated Interferon Alfa-2a; Drug: Highly Active Antiretroviral Therapy (HAART)

INTERVENTIONS:
Drug: Telaprevir — Tablet
  Other Names: VX-950
Drug: Ribavirin — Tablet
  Other Names: Copegus®; RBV
Biological: Pegylated Interferon Alfa-2a — Subcutaneous Injection
  Other Names: Pegasys®; Peg-IFN-Alfa-2a
Drug: Highly Active Antiretroviral Therapy (HAART) — Atazanavir/ritonavir (ATV/r) based HAART, Efavirenz (EFV) based HAART, or Raltegravir (RAL) based HAART, as per standard practice. HAART medications were not considered study drugs.

SUMMARY:
The purpose of this study is to treat human immunodeficiency virus (HIV) and Hepatitis C Virus (HCV) co-infected subjects with telaprevir, pegylated interferon alfa-2a (Peg-IFN-alfa-2a), and ribavirin (RBV) to achieve undetectable hepatitis C virus ribonucleic acid (HCV RNA) 12 weeks after the last planned dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have chronic, genotype 1a or 1b, hepatitis C with HCV RNA greater than (>) 1000 international units per milliliter (IU/mL)
* Population A: HCV Pegylated interferon (Peg-IFN)/RBV treatment naive (received no prior HCV therapy)or Peg-IFN/RBV prior treatment with relapse
* Population B: Peg-IFN/RBV prior null or partial responder
* Participants must not have achieved undetectable HCV RNA 24 weeks after the last planned dose of study drug (SVR24) after at least 1 prior course of Peg IFN/RBV therapy of standard duration
* Participant must have positive HIV antibody at Screening
* Participant must have a diagnosis of HIV-1 infection >6 months before Screening
* Participants should be taking 1 of the following permissible highly active antiretroviral therapy (HAART) regimens for HIV continuously for 12 weeks prior to screening:

  * Atripla® or equivalent components (efavirenz, tenofovir, emtricitabine)
  * Efavirenz plus Epzicom® (abacavir, lamivudine) or equivalent components
  * Boosted atazanavir (atazanavir with ritonavir) plus Truvada® (tenofovir, emtricitabine) or equivalent components
  * Boosted atazanavir plus Epzicom®, or equivalent components
  * Raltegravir plus Truvada®, or equivalent components
  * Raltegravir plus Epzicom®, or equivalent components
* Cluster of differentiation 4 (CD4) counts and human immunodeficiency virus Type 1 (HIV-1) ribonucleic acid (RNA) meeting acceptable criteria at Screening as specified in the protocol
* Laboratory values within acceptable ranges at Screening as specified in the protocol

Exclusion Criteria:

* Subjects anticipating a need to switch HAART regimens within 14 weeks after Day 1 or any switches occurring 12 weeks prior to Day 1
* Use of azidothymidine (AZT), didanosine (ddI) or stavudine (d4T) nucleosides
* Contraindications to any planned HAART component as per the respective drug labeling information
* Contraindications to Peg-IFN or RBV
* Evidence of hepatic decompensation
* Clinical suspicion of acute hepatitis
* Any other cause of liver disease in addition to hepatitis C
* History of organ transplantation (except cornea and skin)
* Autoimmune-mediated disease
* Participated in any investigational drug study within 90 days before Day 1
* Previous treatment with an HCV protease inhibitor

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (59):
- United States (46):
  - Alabama, Birmingham, Alabama
  - California, Bakersfield, California
  - California, Beverly Hills, California
  - California, Coronado, California
  - California, Los Angeles, California
  - California, Oakland, California
  - California, Palo Alto, California
  - California, Sacremento, California
  - California, San Diego, California
  - California, San Francisco, California
  - Connecticut, New Haven, Connecticut
  - DC, Washington D.C., District of Columbia
  - Washington, DC, Washington D.C., District of Columbia
  - Florida, Bay Pines, Florida
  - Florida, Jacksonville, Florida
  - Florida, Miami, Florida
  - Florida, Orlando, Florida
  - Florida, West Palm Beach, Florida
  - Georgia, Atlanta, Georgia
  - Georgia, Decatur, Georgia
  - Illinois, Chicago, Illinois
  - Maine, Portland, Maine
  - Maryland, Baltimore, Maryland
  - Maryland, Lutherville, Maryland
  - Massachusetts, Springfield, Massachusetts
  - Michigan, Detroit, Michigan
  - Minnesota, Minneapolis, Minnesota
  - Missouri, Kansas City, Missouri
  - Missouri, St Louis, Missouri
  - New Jersey, Newark, New Jersey
  - New Mexico, Santa Fe, New Mexico
  - New York, New York, New York
  - New York, Rochester, New York
  - New York, The Bronx, New York
  - North Carolina, Durham, North Carolina
  - Ohio, Cincinnati, Ohio
  - Ohio, Cleveland, Ohio
  - Oregon, Portland, Oregon
  - Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island, Providence, Rhode Island
  - South Carlonia, Columbia, South Carolina
  - Texas, Dallas, Texas
  - Texas, Houston, Texas
  - Utah, Salt Lake City, Utah
  - Virginia, Richmond, Virginia
  - Washington, Seattle, Washington
- Canada (5):
  - Edmonton, Edmonton, Alberta
  - Vancouver, Vancouver, British Columbia
  - Hamilton, Hamilton, Ontario
  - Toronto, Toronto, Ontario
  - Montreal, Montreal, Quebec
- Germany (4):
  - Bonn, Bonn
  - Essen, Essen
  - Hamburg, Hamburg
  - Munchen, München
- Puerto Rico, San Juan, Puerto Rico
- Spain (3):
  - Spain, Badalona
  - Barcelona, Barcelona
  - Madrid, Madrid

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study included Treatment-Naïve (no prior hepatitis C virus [HCV] therapy); Prior Relapser (prior HCV treatment with pegylated interferon alfa/ribavirin [Peg-IFN/RBV] and experienced viral relapse); and Prior Null/Partial Responder (prior HCV treatment with Peg-IFN/RBV and had null/partial response) participants.
Pre-assignment Details: Efficacy analyses were reported as per highly active antiretroviral therapy (HAART) treatment (reporting arms) and also separately as per prior response (in categories) (Treatment-Naive, Prior Relapser, Prior Null Responder, Prior Partial Responder as well as for Total Participants), unless otherwise specified.
Groups:
- T/PR + HAART Regimen (ATV/r-Based): Participants who were receiving atazanavir/ritonavir (ATV/r) based HAART at baseline, received Telaprevir (T)1125 milligram (mg) tablet twice daily for 12 weeks in combination with pegylated interferon alfa 2a (P) (Peg-IFN-alfa-2a) 180 microgram per week (mcg/week) subcutaneous injection and ribavirin (R) (RBV) tablet orally twice daily at a dose of 800 milligram per day (mg/day) for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
- T/PR + HAART Regimen (EFV-Based): Participants who were receiving efavirenz (EFV) based HAART at baseline, received Telaprevir 1125 mg tablet three times a day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 800 mg/day for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
- T/PR + HAART Regimen (RAL-Based): Participants who were receiving raltegravir (RAL) based HAART at baseline, received Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 800 mg/day for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
Period: Overall Study
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Started | 55 | 69 | 61
Treated | 54 | 69 | 59
Completed | 46 | 52 | 45
Not Completed | 9 | 17 | 16
Not completed — No Study Medication | 1 | 0 | 2
Not completed — Adverse Event | 1 | 2 | 0
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Withdrawal of Consent | 3 | 7 | 7
Not completed — Study Terminated by Sponsor | 1 | 3 | 3
Not completed — Other | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS), included all randomized participants who received at least 1 dose of study drug.
Groups:
- T/PR + HAART Regimen (ATV/r-Based): Participants who were receiving ATV/r based HAART at baseline, received Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 800 mg/day for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
- T/PR + HAART Regimen (EFV-Based): Participants who were receiving EFV based HAART at baseline, received Telaprevir 1125 mg tablet three times a day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 800 mg/day for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
- T/PR + HAART Regimen (RAL-Based): Participants who were receiving RAL based HAART at baseline, received Telaprevir 1125 mg tablet twice daily for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 800 mg/day for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their HAART, as per standard practice and investigator discretion.
- Total: Total of all reporting groups
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based) | Total
Number analyzed (Participants) | 54 | 69 | 59 | 182
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.4 (8.81) | 49.6 (8.84) | 48.4 (9.58) | 49.5 (9.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 15 | 30
  Male | 48 | 60 | 44 | 152

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Viral Response 12 Weeks After Last Planned Dose of Study Drug (SVR12)
Description: SVR 12 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (<lower limit of quantification) at 12 weeks after last planned dose of study drug. The plasma hepatitis C virus ribonucleic acid (HCV RNA) level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL).
Time Frame: 12 weeks after last planned dose of study drug (up to Week 60)
Population: Safety Set included all participants who received at least 1 dose of study drug. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 54 | 69 | 59
percentage of participants
  Treatment Naïve (n= 24, 39, 31) | 66.7 | 59.0 | 61.3
  Prior Relapser (n=8, 11, 4) | 75.0 | 54.5 | 100
  Prior Null Responder (n= 15, 11, 15) | 40 | 36.4 | 40
  Prior Partial Responder (n= 7, 8, 9) | 14.3 | 87.5 | 55.6
  Total (n= 54, 69, 59) | 53.7 | 58.0 | 57.6

2. Secondary Outcome: Percentage of Participants With Sustained Viral Response 24 Weeks After Last Planned Dose of Study Drug (SVR 24)
Description: SVR 24 was defined as an undetectable Hepatitis C Virus (HCV) Ribonucleic Acid (RNA) Levels (<lower limit of quantification) at 24 weeks after last planned dose of study drug. The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 international units per milliliter (IU/mL).
Time Frame: 24 weeks after last planned dose of study drug (up to Week 72)
Population: Safety set. Here number of participants analyzed = participants evaluable for this measure and n = participants evaluable for specified categories, for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 53 | 66 | 56
percentage of participants
  Treatment Naïve (n= 23, 38, 29) | 65.2 | 57.9 | 51.7
  Prior Relapser (n=8, 11, 4) | 75.0 | 54.5 | 100
  Prior Null Responder (n= 15, 9, 14) | 33.3 | 22.2 | 35.7
  Prior Partial Responder (n= 7, 8, 9) | 14.3 | 75.0 | 55.6
  Total (n= 53, 66, 56) | 50.9 | 54.5 | 51.8

3. Secondary Outcome: Percentage of Participants With Rapid Viral Response (RVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. RVR was defined as undetectable HCV RNA (<lower limit of quantification) 4 weeks after the start of study treatment.
Time Frame: Week 4
Population: Safety set. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 54 | 69 | 59
percentage of participants
  Treatment Naïve (n= 24, 39, 31) | 50.0 | 53.8 | 74.2
  Prior Relapser (n=8, 11, 4) | 62.5 | 72.7 | 100
  Prior Null Responder (n= 15, 11, 15) | 26.7 | 54.5 | 53.3
  Prior Partial Responder (n= 7, 8, 9) | 42.9 | 50.0 | 44.4
  Total (n= 54, 69, 59) | 44.4 | 56.5 | 66.1

4. Secondary Outcome: Percentage of Participants With Extended Rapid Viral Response (eRVR)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. eRVR was defined as undetectable HCV RNA (<lower limit of quantification) at both 4 weeks and 12 weeks after the start of study treatment.
Time Frame: Week 4 and Week 12
Population: Safety set. Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 54 | 69 | 59
percentage of participants
  Treatment Naïve (n= 24, 39, 31) | 50.0 | 53.8 | 61.3
  Prior Relapser (n=8, 11, 4) | 62.5 | 72.7 | 100
  Prior Null Responder (n= 15, 11, 15) | 26.7 | 54.5 | 53.3
  Prior Partial Responder (n= 7, 8, 9) | 14.3 | 50.0 | 44.4
  Total (n= 54, 69, 59) | 40.7 | 56.5 | 59.3

5. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA at End of Treatment (EOT)
Description: The plasma HCV RNA level was measured using Roche TaqMan HCV RNA assay. The lower limit of quantification was 25 IU/mL. Percentage of participants with undetectable HCV RNA (<lower limit of quantification) at EOT (up to Week 48) are reported. Data for this outcome was not planned to be reported by prior response.
Time Frame: EOT (up to Week 48)
Population: Full analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 54 | 69 | 59
percentage of participants | 55.6 | 63.8 | 61.0

6. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE: any untoward medical occurrence in a participant during the study; the event does not necessarily have a causal relationship with the treatment. This includes any newly occurring event or previous condition that has increased in severity or frequency after the informed consent form is signed. SAE (subset of AE): medical event or condition, which falls into any of the following categories, regardless of its relationship to the study drug: death, life threatening adverse experience, in-patient hospitalization/prolongation of hospitalization, persistent/significant disability or incapacity, congenital anomaly/birth defect, important medical event.
Time Frame: Up to Week 52
Population: Safety set.
Measure: Number; unit: percentage of participants
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 54 | 69 | 59
percentage of participants
  AEs | 100 | 95.7 | 94.9
  SAEs | 13.0 | 11.6 | 15.3

7. Secondary Outcome: Maximum (Cmax), Minimum (Cmin), and Average Plasma Concentration (Cavg)
Description: Cmax, Cmin, and Cavg were reported for atazanavir (ATV), efavirenz (EFV), raltegravir (RAL), and telaprevir.
Time Frame: Day -14 to Day -1 and Week 1 for ATV, EFV, and RAL; Week 1 for telaprevir
Population: Full Analysis set.Here, n = participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Number analyzed (Participants) | 54 | 69 | 59
nanogram per milliliter (ng/mL)
  ATV: Day -14 to Day -1, Cmax(n=46, 0, 0) | 2870 (1580) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  ATV: Day -14 to Day -1, Cmin(n=46, 0, 0) | 991 (635) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  ATV: Day -14 to Day -1, Cavg(n=41, 0, 0) | 1100 (647) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  ATV: Week 1, Cmax (n=42, 0, 0) | 2820 (1570) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  ATV: Week 1, Cmin (n=42, 0, 0) | 1280 (636) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  ATV: Week 1, Cavg (n=30, 0, 0) | 1320 (685) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  EFV: Day -14 to Day -1, Cmax(n=0, 60, 0) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 3800 (2600) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  EFV: Day -14 to Day -1, Cmin(n=0, 60, 0) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 2560 (1900) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  EFV: Day -14 to Day -1, Cavg(n=0, 51, 0) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 2150 (1680) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  EFV: Week 1, Cmax (n=0, 51, 0) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 3340 (2450) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  EFV: Week 1, Cmin (n=0, 51, 0) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 2290 (1880) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  EFV: Week 1, Cavg (n=0, 47, 0) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 1920 (1400) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group
  RAL: Day -14 to Day -1, Cmax(n=0, 0, 52) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 1900 (1880)
  RAL: Day -14 to Day -1, Cmin(n=0, 0, 52) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 196 (198)
  RAL: Day -14 to Day -1, Cavg(n=0, 0, 35) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 483 (429)
  RAL: Week 1, Cmax (n=0, 0, 49) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 2320 (1970)
  RAL: Week 1, Cmin (n=0, 0, 49) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 281 (435)
  RAL: Week 1, Cavg (n=0, 0, 34) | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | NA (NA) — Data not reported as no participant was evaluable for this parameter from this reporting group | 643 (539)
  Telaprevir: Week 1, Cmax(n=49, 59, 54) | 3160 (1180) | 3780 (1670) | 3470 (868)
  Telaprevir: Week 1, Cmin(n=49, 59, 54) | 1650 (863) | 1750 (961) | 1840 (741)
  Telaprevir: Week 1, Cavg(n=30, 32, 26) | 2320 (907) | 2430 (1290) | 2520 (643)

8. Secondary Outcome: Number of Participants With Telaprevir Resistant HCV Variant at Non-Structural Viral Protein 3-4A (NS3-4A) Region
Description: Sequence analysis of the HCV NS3-4A region was performed to monitor telaprevir-resistant variants. HCV RNA was isolated from the plasma, amplified by reverse transcription-polymerase chain reaction (RT-PCR), and sequenced (sequencing assay limit of detection HCV RNA >=1000 IU/mL). Results of this outcome measure were to be reported for overall participants instead of by HAART treatment.
Time Frame: Baseline, follow-up (Week 96)
Population: Full analysis set. Here number of participants analyzed = participants who were evaluable for this measure and n = participants evaluable for specified categories.
Measure: Number; unit: participants
Groups:
- T/PR + HAART Regimen: Participants who were receiving either ATV/r based HAART or EFV based HAART or RAL based HAART at baseline, received Telaprevir 1125 mg tablet twice daily or 1125 mg three times a day for 12 weeks in combination with Peg-IFN-alfa-2a 180 mcg/week subcutaneous injection and RBV tablet orally twice daily at a dose of 800 mg/day for 24 or 48 weeks, depending on individual response to telaprevir treatment. Participants continued their respective HAART, as per standard practice and investigator discretion.
Arm/Group | T/PR + HAART Regimen
Number analyzed (Participants) | 180
participants
  Baseline (n = 180) | 2
  Follow-up (n = 26) | 11

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: Adverse events were planned to be reported as per HAART treatment.
Arm/Group | T/PR + HAART Regimen (ATV/r-Based) | T/PR + HAART Regimen (EFV-Based) | T/PR + HAART Regimen (RAL-Based)
Serious Adverse Events (participants affected / at risk) | 7/54 | 8/69 | 9/59
Other Adverse Events (participants affected / at risk) | 54/54 | 66/69 | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T/PR + HAART Regimen (ATV/r-Based) (N=54) | T/PR + HAART Regimen (EFV-Based) (N=69) | T/PR + HAART Regimen (RAL-Based) (N=59)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 4
Neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Psoas abscess (Infections and infestations) | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 0 | 1
Retinopathy (Eye disorders) | 0 | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | T/PR + HAART Regimen (ATV/r-Based) (N=54) | T/PR + HAART Regimen (EFV-Based) (N=69) | T/PR + HAART Regimen (RAL-Based) (N=59)
Nausea (Gastrointestinal disorders) | 23 (27) | 22 (26) | 19 (23)
Diarrhoea (Gastrointestinal disorders) | 13 (14) | 21 (22) | 6 (6)
Vomiting (Gastrointestinal disorders) | 10 (10) | 11 (14) | 11 (15)
Anorectal discomfort (Gastrointestinal disorders) | 6 (6) | 11 (11) | 9 (10)
Anal pruritus (Gastrointestinal disorders) | 4 (4) | 10 (10) | 6 (6)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 11 (11) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1) | 5 (5)
Constipation (Gastrointestinal disorders) | 2 (2) | 5 (5) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 3 (3)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Flatulence (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (2) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Loose tooth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abnormal faeces (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anorectal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dental caries (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal tract irritation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral mucosal erythema (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Palatal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue eruption (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 26 (32) | 36 (43) | 30 (34)
Influenza like illness (General disorders) | 5 (5) | 8 (9) | 8 (8)
Pyrexia (General disorders) | 9 (10) | 5 (5) | 7 (7)
Chills (General disorders) | 8 (8) | 6 (6) | 4 (5)
Asthenia (General disorders) | 6 (6) | 2 (2) | 9 (9)
Injection site reaction (General disorders) | 1 (1) | 9 (9) | 4 (4)
Irritability (General disorders) | 2 (2) | 5 (6) | 7 (8)
Pain (General disorders) | 6 (6) | 2 (2) | 6 (6)
Injection site erythema (General disorders) | 0 (0) | 3 (5) | 2 (2)
Malaise (General disorders) | 0 (0) | 2 (3) | 2 (2)
Injection site bruising (General disorders) | 0 (0) | 2 (2) | 1 (1)
Injection site rash (General disorders) | 0 (0) | 1 (1) | 2 (2)
Crying (General disorders) | 0 (0) | 1 (1) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 2 (2) | 0 (0)
Thirst (General disorders) | 1 (1) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cyst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Feeling abnormal (General disorders) | 0 (0) | 1 (1) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 0 (0) | 1 (1)
Local swelling (General disorders) | 0 (0) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0)
Sluggishness (General disorders) | 0 (0) | 1 (1) | 0 (0)
Temperature intolerance (General disorders) | 0 (0) | 1 (1) | 0 (0)
Xerosis (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 22 (25) | 21 (22) | 18 (20)
Rash (Skin and subcutaneous tissue disorders) | 16 (23) | 20 (25) | 11 (15)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 4 (4)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (4) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash morbilliform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Skin fissures (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 15 (17) | 17 (18) | 20 (23)
Dizziness (Nervous system disorders) | 6 (7) | 6 (6) | 6 (7)
Dysgeusia (Nervous system disorders) | 2 (2) | 10 (10) | 5 (5)
Disturbance in attention (Nervous system disorders) | 0 (0) | 4 (4) | 4 (4)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 4 (5)
Dizziness postural (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 2 (5) | 1 (1)
Hypersomnia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Allodynia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sensory disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 15 (17) | 21 (23) | 16 (20)
Neutropenia (Blood and lymphatic system disorders) | 10 (13) | 15 (23) | 4 (6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 5 (6) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Lymphoid tissue hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 9 (9) | 14 (15) | 14 (16)
Depression (Psychiatric disorders) | 5 (6) | 7 (8) | 4 (4)
Mood swings (Psychiatric disorders) | 2 (2) | 5 (5) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (3) | 2 (2)
Sleep disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (3)
Affect lability (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Bruxism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Libido decreased (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Mood altered (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Stress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (9) | 9 (9)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 5 (7)
Folliculitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (2) | 2 (2) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Oral candidiasis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (2)
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Onychomycosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Abscess jaw (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Abscess soft tissue (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Cardiac valve vegetation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Injection site pustule (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mycoplasma infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethritis chlamydial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urethritis gonococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (9) | 11 (12) | 8 (8)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 6 (6) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (4) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Abnormal loss of weight (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperlipasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (5) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Increased viscosity of nasal secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal plaque (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 3 (3) | 6 (6) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 3 (3)
Blood uric acid increased (Investigations) | 1 (1) | 1 (1) | 2 (3)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (2) | 0 (0) | 1 (2)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood triglycerides increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eosinophil count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haematocrit decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Prothrombin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Reticulocyte count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1) | 1 (1)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Visual impairment (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Abnormal sensation in eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis allergic (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Eye discharge (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye inflammation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Hypermetropia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Ocular icterus (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block first degree (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Pyuria (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Enuresis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Genital hypoaesthesia (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Menstruation irregular (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Jaundice (Hepatobiliary disorders) | 3 (3) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0) | 1 (1)
Hypogonadism (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Colour blindness (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0)
Seasonal allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
It was decided by Sponsor on 13 January 2014 to terminate the study early at the primary efficacy endpoint (SVR12) as part of a decision to modify the drug development plan. Eligible participants completed virologic follow-up after termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI is free to publish results of the study after (1) the first multi-center publication, (2) if the sponsor elects not to publish the results, or (3) 18 months after close of the study, whichever occurs first. Proposed publications are to be submitted to the sponsor for review and comment for a period of at least 45 days (which may be extended under certain circumstances related to protection of intellectual property); the sponsor cannot require changes to the proposed publications.